CLINICAL TRIAL: NCT00812448
Title: The Effects of Tea Catechin Extracts Containing Mask on the Prevention of Influenza Infection
Brief Title: Catechin Containing Mask for the Prevention of Influenza Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Shizuoka (Other)
Collaborators: Seirei Hamamatsu General Hospital (Other); Hamamatsu University (Other)
Responsible Party: Hiroshi Yamada/Professor, University of Shizuoka
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CT2009001; 20-24
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Last update posted 2009-11-26 (Estimated); Status verified 2009-11

CONDITIONS: Influenza Infection
Keywords: prophylaxis; influenza infection; catechins; prophylaxis of influenza infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tea catechin extracts containing mask (Experimental): wearing the tea catechin extracts containing mask
  Interventions: Dietary Supplement: tea catechin extracts

INTERVENTIONS:
Dietary Supplement: tea catechin extracts — catechins are composed of tea catechin extracts available in grren tea supplements

SUMMARY:
The purpose of this study is to evaluate the effects of catechin extracts containing mask on prevention of influenza infection.

DETAILED DESCRIPTION:
Catechins are the major components of tea flavonoids and are reported to possess physiological activities such as antiviral effects. Recent in-vitro experimental studies have revealed that tea catechin extracts possess the effects on the prevention of influenza infection. However, a limited number of studies have been conducted on the clinical effects. Based on these backgrounds, we designed a prospective randomized controlled study to evaluate the effects of tea catechin extracts containing mask on the prevention of influenza infection.

ELIGIBILITY:
Inclusion Criteria:

* Possible to wearing mask for three months
* Possible to fill out a questionnaire personally
* Obtained written informed consent before participation

Exclusion Criteria:

* Possessing some infectious diseases in need of therapy
* Possessing tea or catechin allergy
* diagnosed as inadequate for other reasons to participate the study by principal investigator

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2008-12; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
the incidence rate of influenza infection during the study | assessed at each month

SECONDARY OUTCOMES:
the incidence rates of upper respiratory tract infections | assessed at each month
the severity of the symptoms and the duration of the cold among incident cases | assessed at each month
he incidence-free time for influenza or upper respiratory tract infections after the intervention | assessed at each month

CONTACTS AND LOCATIONS:
Overall Officials: Hiroshi Yamada, MD,PhD, Study Chair — University of Shizuoka
Locations (2):
- Japan (2):
  - Seirei Hamamatsu General Hospital, Hamamatsu, Shizuoka
  - University of Shizuoka, Shizuoka, Shizuoka